CLINICAL TRIAL: NCT00542152
Title: A Randomized, Multicenter Open Label Study Comparing Cyclosporine With Infliximab in Steroid-refractory Severe Attacks of Ulcerative Colitis
Brief Title: Study Comparing Cyclosporine With Infliximab in Steroid-refractory Severe Attacks of Ulcerative Colitis
Acronym: CYSIF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2006-3
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Ulcerative Colitis; Steroid Refractory
Keywords: IBD; Ulcerative colitis; refractory to steroids
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Cyclosporine; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CICLO (Active Comparator): Cyclosporine will be administered by continuous intravenous infusion at the initial dose regimen of 2mg/kg per day.
  After 24 hours of treatment, cyclosporine trough level will be measured and the dose adapted in order to obtain a cyclosporinaemia level between 150 and 250 ng/ml. Cyclosporinaemia will be reassessed every 48 hours for the duration of the continuous intravenous treatment.
  Interventions: Drug: CYCLOSPORINE VS INFLIXIMAB
- INFLIXIMAB (Active Comparator): INFLIXIMAB (REMICADE) Infliximab in the form of a freeze-dried compound is conditioned in 100mg vials. Treatment will first be reconstituted in 250ml isotonic saline solution, and slowly infused at the dose of 5mg/kg in 2 hours.
  In patients with clinical response at D7 (Lichtiger Index score < 10 for 2 consecutive days), two additional infliximab infusions will be administered at the dose of 5mg/kg at D14 and D42.
  Interventions: Drug: CYCLOSPORINE VS INFLIXIMAB

INTERVENTIONS:
Drug: CYCLOSPORINE VS INFLIXIMAB — * Cyclosporine 2mg/kg/day intravenous for 7 days then Neoral 4mg/kg/day orally for 3 months.
  * Infliximab 5mg/kg at weeks 0, 2 and 6
  Other Names: Cyclosporine (IV)= Brand Name = Sandinuum; Cyclosporine (PO)= brand name = Neoral; Infliximab (IV)= brand name= Remicade

SUMMARY:
PHASE: IV

TYPE OF STUDY: With direct benefit.

DESCRIPTIVE: Multicenter, randomized, open label study.

INCLUSION CRITERIA: Steroid-refractory ulcerative colitis.

OBJECTIVES: To compare the efficacy of cyclosporine with infliximab in steroid- refractory attacks of ulcerative colitis.

STUDY TREATMENTS:Cyclosporine 2mg/kg/day intravenous(IV)for 7days then Neoral 4mg/kg/day orally for 3 months. Infliximab 5mg/kg at Weeks 0, 2 and 6.

NUMBER OF PATIENTS: 50 patients in each group i.e. a total of 100 patients.

INCLUSION PERIOD: 24 months.

STUDY DURATION: 27 months.

MAIN EVALUATION CRITERIA:

Clinical response at D7 according to the Lichtiger Index score AND Clinical Remission at D98 according to the Mayo Disease Activity Index score

SECONDARY EVALUATION CRITERIA:

Clinical remission at D98 (according to the Mayo Disease Activity Index score) Endoscopic response Colectomy rate Tolerance

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Diagnosis of UC according to Lennard-Jones criteria (Appendix 1).
* Endoscopically demonstrated colorectal lesions localized above the anal margin and extending at least up to 15cm proximally.
* Severe acute flare of UC with a Lichtiger Index score > 10.
* Refractoriness to high dose intravenous steroid therapy (≥ 0.8 mg/kg/d of methylprednisolone or equivalent) given for at least 5 days.
* Adequate contraception for male or female subjects of childbearing potential, which will be continued throughout the study and at least 3 months after study termination.

Exclusion Criteria:

* Pregnant or breast-feeding woman.
* Previous treatment with cyclosporine or infliximab.
* Azathioprine or 6-mercaptopurine treatment initiated more than 4 weeks before inclusion.
* Indication for immediate surgery.
* History of colorectal dysplasia.
* Diagnosis of Crohn's disease.
* Positive stool tests for amoebiasis and/or positive bacteriological culture for Salmonella, Shigella, Yersinia and Campylobacter and/or presence of Clostridium difficile B toxin in the stools.
* Renal failure (creatininemia > upper limit of normal laboratory value).
* Uncontrolled high blood pressure.
* HIV, HBV viral infection (except the presence of positive anti-HBs antibodies) with serology not older than 3 months.
* Uncontrolled bacterial or active viral infection.
* Past medical history of malignant condition in the last 5 years (including leukaemia, lymphoma and myelodysplasia) except for baso-cellular cutaneous cancers.
* Past medical history of myocardial infarction or heart failure.
* Intradermal reaction to Tuberculin (Tubertest® 5 units) > 5mm.
* Active tuberculosis
* Untreated latent tuberculosis (see national recommendations. Appendix 2).
* Abnormal blood count with polynuclear neutrophils < 1,500 G/L or white cells < 3,000, or platelets < 100,000 G/L.
* Unexplained rise higher than 3 times the normal level for transaminases, alkaline phosphatases and/or higher than twice the normal level for bilirubin.
* Non-compliant subjects.
* Participation in another therapeutic study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-06; Primary Completion 2007-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
% of patients with treatment failure defined as: absence of clinical response at D7 or absence of remission without steroids at D98 or relapse or severe adverse event leading to treatment interruption or colectomy or fatality between D0 and D98 | Day 7

SECONDARY OUTCOMES:
% of patients in clinical response % patients in remission Lichtiger Index score MDAI score Time to discharge Endoscopic response colectomy rate Steroid dosage. Number of adverse events CMV infection | D98

CONTACTS AND LOCATIONS:
Overall Officials: David LAHARIE, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (41):
- Belgium (4):
  - Hopital Erasme, Brussels
  - Ulb - Clinique Saint Luc, Brussels
  - Gent University Hospital, Ghent
  - Leuven University Hospital, Leuven
- Helsinki University Hospital, Helsinki, Finland
- France (31):
  - Chu Amiens, Amiens
  - Ch Avignon, Avignon
  - Chu Besancon, Besançon
  - CHU CAEN, Caen
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Louis Mourrier, Colombes
  - Hopital Henri Mondor, Créteil
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Chru Lille, Lille
  - Chu Marseille - Hopital Nord, Marseille
  - Ch Le Raincy Montfermeil, Montfermeil
  - Chu Nantes, Nantes
  - CHU NICE, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Saint Louis, Paris
  - Hopital St Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Georges Pompidou, Paris
  - Hopital Bichat, Paris
  - Institut Mutualiste Montsouris (Imm), Paris
  - Hopital Haut Leveque, Pessac
  - CHU LYON, Pierre-Bénite
  - Chu Reims, Reims
  - Chu Rennes, Rennes
  - Chu Rouen, Rouen
  - Chu Saint Etienne, Saint-Etienne
  - Chu Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - Chu Tours, Tours
  - Chu Nancy, Vandœuvre-lès-Nancy
- Istituto Clinico Humanitas, Milan, Italy
- Spain (4):
  - Hospital Clinic, Barcelona
  - Hospital Mutua de Terressa, Barcelona
  - Hospital de la Princesa, Madrid
  - Hospital Ramon Y Cajal, Madrid

REFERENCES:
- [Background] EDWARDS FC, TRUELOVE SC. THE COURSE AND PROGNOSIS OF ULCERATIVE COLITIS. Gut. 1963 Dec;4(4):299-315. doi: 10.1136/gut.4.4.299. PMID 14084741
- [Background] Truelove SC, Willoughby CP, Lee EG, Kettlewell MG. Further experience in the treatment of severe attacks of ulcerative colitis. Lancet. 1978 Nov 18;2(8099):1086-8. doi: 10.1016/s0140-6736(78)91816-0. PMID 82099
- [Background] D'Haens G, Lemmens L, Geboes K, Vandeputte L, Van Acker F, Mortelmans L, Peeters M, Vermeire S, Penninckx F, Nevens F, Hiele M, Rutgeerts P. Intravenous cyclosporine versus intravenous corticosteroids as single therapy for severe attacks of ulcerative colitis. Gastroenterology. 2001 May;120(6):1323-9. doi: 10.1053/gast.2001.23983. PMID 11313301
- [Background] Lichtiger S, Present DH, Kornbluth A, Gelernt I, Bauer J, Galler G, Michelassi F, Hanauer S. Cyclosporine in severe ulcerative colitis refractory to steroid therapy. N Engl J Med. 1994 Jun 30;330(26):1841-5. doi: 10.1056/NEJM199406303302601. PMID 8196726
- [Background] Van Assche G, D'Haens G, Noman M, Vermeire S, Hiele M, Asnong K, Arts J, D'Hoore A, Penninckx F, Rutgeerts P. Randomized, double-blind comparison of 4 mg/kg versus 2 mg/kg intravenous cyclosporine in severe ulcerative colitis. Gastroenterology. 2003 Oct;125(4):1025-31. doi: 10.1016/s0016-5085(03)01214-9. PMID 14517785
- [Background] Arts J, D'Haens G, Zeegers M, Van Assche G, Hiele M, D'Hoore A, Penninckx F, Vermeire S, Rutgeerts P. Long-term outcome of treatment with intravenous cyclosporin in patients with severe ulcerative colitis. Inflamm Bowel Dis. 2004 Mar;10(2):73-8. doi: 10.1097/00054725-200403000-00002. PMID 15168804
- [Background] Actis GC, Bresso F, Astegiano M, Demarchi B, Sapone N, Boscaglia C, Rizzetto M. Safety and efficacy of azathioprine in the maintenance of ciclosporin-induced remission of ulcerative colitis. Aliment Pharmacol Ther. 2001 Sep;15(9):1307-11. doi: 10.1046/j.1365-2036.2001.01019.x. PMID 11552900
- [Background] Cohen RD, Stein R, Hanauer SB. Intravenous cyclosporin in ulcerative colitis: a five-year experience. Am J Gastroenterol. 1999 Jun;94(6):1587-92. doi: 10.1111/j.1572-0241.1999.01149.x. PMID 10364029
- [Background] Ardizzone S, Maconi G, Russo A, Imbesi V, Colombo E, Bianchi Porro G. Randomised controlled trial of azathioprine and 5-aminosalicylic acid for treatment of steroid dependent ulcerative colitis. Gut. 2006 Jan;55(1):47-53. doi: 10.1136/gut.2005.068809. Epub 2005 Jun 21. PMID 15972298
- [Background] Shibolet O, Regushevskaya E, Brezis M, Soares-Weiser K. Cyclosporine A for induction of remission in severe ulcerative colitis. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD004277. doi: 10.1002/14651858.CD004277.pub2. PMID 15674937
- [Background] Jarnerot G, Hertervig E, Friis-Liby I, Blomquist L, Karlen P, Granno C, Vilien M, Strom M, Danielsson A, Verbaan H, Hellstrom PM, Magnuson A, Curman B. Infliximab as rescue therapy in severe to moderately severe ulcerative colitis: a randomized, placebo-controlled study. Gastroenterology. 2005 Jun;128(7):1805-11. doi: 10.1053/j.gastro.2005.03.003. PMID 15940615
- [Background] Su C, Salzberg BA, Lewis JD, Deren JJ, Kornbluth A, Katzka DA, Stein RB, Adler DR, Lichtenstein GR. Efficacy of anti-tumor necrosis factor therapy in patients with ulcerative colitis. Am J Gastroenterol. 2002 Oct;97(10):2577-84. doi: 10.1111/j.1572-0241.2002.06026.x. PMID 12385442
- [Background] Gornet JM, Couve S, Hassani Z, Delchier JC, Marteau P, Cosnes J, Bouhnik Y, Dupas JL, Modigliani R, Taillard F, Lemann M. Infliximab for refractory ulcerative colitis or indeterminate colitis: an open-label multicentre study. Aliment Pharmacol Ther. 2003 Jul 15;18(2):175-81. doi: 10.1046/j.1365-2036.2003.01686.x. PMID 12869077
- [Background] Kohn A, Prantera C, Pera A, Cosintino R, Sostegni R, Daperno M. Infliximab in the treatment of severe ulcerative colitis: a follow-up study. Eur Rev Med Pharmacol Sci. 2004 Sep-Oct;8(5):235-7. PMID 15638237
- [Background] Eidelwein AP, Cuffari C, Abadom V, Oliva-Hemker M. Infliximab efficacy in pediatric ulcerative colitis. Inflamm Bowel Dis. 2005 Mar;11(3):213-8. doi: 10.1097/01.mib.0000160803.44449.a5. PMID 15735427
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Derived] Hasskamp J, Meinhardt C, Patton PH, Timmer A. Azathioprine and 6-mercaptopurine for maintenance of remission in ulcerative colitis. Cochrane Database Syst Rev. 2025 Feb 27;2(2):CD000478. doi: 10.1002/14651858.CD000478.pub5. PMID 40013523
- [Derived] Laharie D, Bourreille A, Branche J, Allez M, Bouhnik Y, Filippi J, Zerbib F, Savoye G, Vuitton L, Moreau J, Amiot A, Cosnes J, Ricart E, Dewit O, Lopez-Sanroman A, Fumery M, Carbonnel F, Bommelaer G, Coffin B, Roblin X, van Assche G, Esteve M, Farkkila M, Gisbert JP, Marteau P, Nahon S, de Vos M, Lambert J, Mary JY, Louis E; Groupe d'Etudes Therapeutiques des Affections Inflammatoires Digestives. Long-term outcome of patients with steroid-refractory acute severe UC treated with ciclosporin or infliximab. Gut. 2018 Feb;67(2):237-243. doi: 10.1136/gutjnl-2016-313060. Epub 2017 Jan 4. PMID 28053054
- [Derived] Laharie D, Bourreille A, Branche J, Allez M, Bouhnik Y, Filippi J, Zerbib F, Savoye G, Nachury M, Moreau J, Delchier JC, Cosnes J, Ricart E, Dewit O, Lopez-Sanroman A, Dupas JL, Carbonnel F, Bommelaer G, Coffin B, Roblin X, Van Assche G, Esteve M, Farkkila M, Gisbert JP, Marteau P, Nahon S, de Vos M, Franchimont D, Mary JY, Colombel JF, Lemann M; Groupe d'Etudes Therapeutiques des Affections Inflammatoires Digestives. Ciclosporin versus infliximab in patients with severe ulcerative colitis refractory to intravenous steroids: a parallel, open-label randomised controlled trial. Lancet. 2012 Dec 1;380(9857):1909-15. doi: 10.1016/S0140-6736(12)61084-8. Epub 2012 Oct 10. PMID 23063316
- See also: Related Info — http://www.getaid.org